CLINICAL TRIAL: NCT04589273
Title: The Effect of Alginate Supplementation on Weight Management - A Randomised Double Blind Placebo Controlled Pilot Trial
Brief Title: The Effect of Alginate Supplementation on Weight Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1882/1283
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Overweight and Obesity
Keywords: obesity; overweight
MeSH Terms: conditions — Overweight; Obesity | interventions — Alginates

STUDY DESIGN:
Intervention Model Description: Double blind, randomised, placebo controlled trial
Who Masked: Participant, Investigator
Masking Description: Neither the researcher or the participant will know which arm of the trial they are part of.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alginate capsule (Experimental): The participants of this arm will be give the alginate capsules
  Interventions: Dietary Supplement: Alginate
- Placebo (Placebo Comparator): The participants of this arm will be give the placebo capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Alginate — Volunteers will be asked to consume the alginate capsules with each of their three main meals per day.
  Arms: Alginate capsule
Other: Placebo — Volunteers will be asked to consume the placebo capsules with each of their three main meals per day.
  Arms: Placebo

SUMMARY:
This project will assess the effect of the alginate (in a capsules) on the weight of generally healthy volunteers over a 12 week period.

To achieve this, will recruit 150 (non-smoking) generally healthy volunteers to attend the study centre on four separate occasions. Volunteers will be randomly allocated into active or placebo arm of the trial, both will receive capsules with the same appearance.

The volunteers will have their height, weight, waist circumference, body composition, and fasting levels of circulating glucose, triacylglycerol and cholesterol measured at each for the four visits.

DETAILED DESCRIPTION:
The study will last approximately 12 weeks depending on your availability.

Volunteers will be asked to come to the research facility in Newcastle University, before they have had any breakfast, on four separate occasions. The volunteers must not eat or drink anything (except water) after 8 pm the evening before they come in. This includes not drinking any alcohol, tea or coffee.

Each time the volunteers come in, their height (first assessment only), weight, waist circumference and body composition will be measured. Body composition is measured using scales which can determine the percentage of their body is fat or bone or muscle. This is done using a small harmless electrical current passing through their body, they will not detect or feel this at all. Their height will also be measured at the first visit. Cholesterol, triglyceride and glucose levels in the blood will also be measured at each visit. This will be done through a single finger prick blood sample.

Enough capsules will be given to the volunteers to last you four weeks at the first three visits. The capsules will be filled with either alginate or another dietary fibre believed to have no effect on weight management.

Volunteers will be asked to take four of these capsules with their three main meals per day over the 12 week study.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* BMI over 20

Exclusion Criteria:

* Pregnant, lactating,
* BMI under 20

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | 12 weeks
  A change in weight measured in kg
Change in amount of body fat | 12 weeks
  A change in body fat (as a percentage) as measured by impedance

SECONDARY OUTCOMES:
Change in waist circumference | 12 weeks
  A change in waist circumference measured in cm
Change in fasting Cholesterol | 12 weeks
  A change in fasting circulating cholesterol
Change in fasting Glucose | 12 weeks
  A Change in fasting circulating glucose
Change in fasting triacylglycerol | 12 weeks
  A change in fasting circulating triacylglycerol

CONTACTS AND LOCATIONS:
Overall Officials: Pearson, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Newcastle, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No